CLINICAL TRIAL: NCT03636958
Title: Study of the Efficacy and Safety of Perampanel in Combination in Glioma-refractory Epilepsy
Brief Title: Efficacy and Safety of Perampanel in Combination in Glioma-refractory Epilepsy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: concomitant decision of the sponsor and the PI, lack of patients
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-13
Record Dates: First submitted 2018-08-16; First posted 2018-08-17 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Refractory Epilepsy
MeSH Terms: conditions — Drug Resistant Epilepsy | interventions — perampanel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): they will receive conventional antiepileptic treatment (antiepileptic combination therapy) without perampanel
  Interventions: Drug: conventional antiepileptic treatment
- experimental group (Experimental): they will receive conventional antiepileptic treatment (antiepileptic combination therapy) with perampanel
  Interventions: Drug: Perampanel; Drug: conventional antiepileptic treatment

INTERVENTIONS:
Drug: Perampanel — Perampanel is an antiepileptic with a novel mechanism of action as it targets post-synaptic AMPA receptors. It has been shown to be effective as adjunctive therapy (dual therapy) for partial / focal epilepsy seizures and generalized in patients over 12 years of age.
  Arms: experimental group
Drug: conventional antiepileptic treatment — choice of the molecule is left to the discretion of the clinician excluding the following benzodiazepines: clobazam, clonazepam, diazepam. Antiepileptic drugs allowed are therefore: lamotrigine, levetiracetam, lacosamide, sodium valproate, carbamazepine, oxcarbabazepine, slicarbazepine, pregabalin, gabapentin, topiramate, phenytoin, phenobarbital, zonisamide, vigabatrin.

SUMMARY:
Gliomas are primitive brain tumors frequently associated with epilepsy. In a significant number of these patients epilepsy is resistant to antiepileptic drugs. There are currently no recommendations for the management of these drug-resistant epilepsies associated with glioma. In addition, few studies have addressed the subject and no treatment appears to be superior to others in the literature for this indication. In addition, many antiepileptic drugs pose problems of tolerance or interaction with chemotherapy in these patients.

Fundamental studies on glioma-associated epilepsies have shown that there is a major dysregulation of glutamatergic systems involved in epileptogenesis and tumor growth. Targeting this glutamatergic system seems particularly interesting from a physiopathological point of view. Perampanel is a recent antiepileptic treatment with a novel mode of action targeting AMPA glutamate receptors. It has been shown to be effective in patients with drug-resistant epilepsies. He has demonstrated his tolerance in these patients. He has obtained a marketing authorization and is therefore used in routine epileptology without serious problems of tolerance being reported. It is neither an inducer nor an enzyme inhibitor, avoiding the problems of interaction with chemotherapy and is used in a daily dose facilitating compliance.

Therefore, there may be specific antiepileptic efficacy of perampanel in patients with glioma. Nevertheless, the only current data is limited to a retrospective study of 12 patients.

The objective of this protocol is to evaluate the efficacy and safety of perampanel in patients with glioma with drug-resistant epilepsy.

a prospective randomized study with two parallel arms: antiepileptic combination therapy with perampanel and antiepileptic combination therapy without perampanel (free choice of the practitioner). The main criterion of judgment will be the decrease of the monthly frequency of crisis. Secondary endpoints will assess tolerance, efficacy on responder rate (at least 50% decrease in seizure frequency), seizure severity (secondary generalization, loss of consciousness), and quality. patients' lives (quality of life questionnaires, side effects and anxiety / depression). The duration of participation per patient will be 23 weeks (6 weeks of baseline, 5 weeks of titration and 12 weeks of maintenance). The recruitment period will be 3 years. Investigators plan to recruit 120 patients.

In the context of no recommendation in the management of these patients, superior efficacy of perampanel compared with other antiepileptic drugs is expected. This would allow targeted treatment in this population and confirm the tolerance of this treatment in these patients.

DETAILED DESCRIPTION:
Background: Gliomas are primitive brain tumors frequently associated with epilepsy. In a significant number of these patients epilepsy is resistant to antiepileptic drugs. There are currently no recommendations for the management of these drug-resistant epilepsies associated with glioma. In addition, few studies have addressed the subject and no treatment appears to be superior to others in the literature for this indication. In addition, many antiepileptic drugs pose problems of tolerance or interaction with chemotherapy in these patients.

Rational: Fundamental studies on glioma-associated epilepsies have shown that there is a major dysregulation of glutamatergic systems involved in epileptogenesis (= perpetuation of epileptic seizures) and tumor growth (Huberfeld and Vecht, 2016). Targeting this glutamatergic system seems particularly interesting from a physiopathological point of view. Perampanel is a recent antiepileptic treatment with a novel mode of action targeting AMPA glutamate receptors. It has been shown to be effective in patients with drug-resistant epilepsies. He has demonstrated his tolerance in these patients. He has obtained a marketing authorization and is therefore used in routine epileptology without serious problems of tolerance being reported. It is neither an inducer nor an enzyme inhibitor, avoiding the problems of interaction with chemotherapy and is used in a daily dose facilitating compliance.

Therefore, there may be specific antiepileptic efficacy of perampanel in patients with glioma. Nevertheless, the only current data is limited to a retrospective study of 12 patients.

The objective of this protocol is to evaluate the efficacy and safety of perampanel in patients with glioma with drug-resistant epilepsy.

The investigators want to perform a prospective randomized study with two parallel arms: antiepileptic combination therapy with perampanel and antiepileptic combination therapy without perampanel (free choice of the practitioner). The main criterion of judgment will be the decrease of the monthly frequency of crisis. Secondary endpoints will assess tolerance, efficacy on responder rate (at least 50% decrease in seizure frequency), seizure severity (secondary generalization, loss of consciousness), and quality. patients' lives (quality of life questionnaires, side effects and anxiety / depression). The duration of participation per patient will be 23 weeks (6 weeks of baseline, 5 weeks of titration and 12 weeks of maintenance). The recruitment period will be 3 years. The investigators plan to recruit 120 patients.

Expected benefits: In the context of no recommendation in the management of these patients, the investigators hope to demonstrate superior efficacy of perampanel compared with other antiepileptic drugs. This would allow targeted treatment in this population and confirm the tolerance of this treatment in these patients.

ELIGIBILITY:
Inclusion Criteria:

Patient, male or female, over 18 years old

* Glioma confirmed by histology
* Not in progression (clinico-radiological criterion RANO, (Wen et al., 2014), see appendix 1)

  * No clinical worsening (excluding epileptic seizures)
  * No increase greater than 25% in contrast enhancement after gadolinium injection
  * No increase in the T2 / FLAIR hyper signal
  * Absence of new lesion
* Diagnosis of drug-resistant epilepsy according to international epilepsy definitions (Fisher 2014 and Kwan 2010, see Appendices 2 and 3)

  o Repeated epileptic seizures despite testing of two effective dose antiepileptic drugs tried at least 3 months
* With at least 2 attacks per month (to ensure visibility on the duration of the study of the antiepileptic effect, see below)
* Patient with epileptic seizures not limited to only subjective signs

Exclusion Criteria:

* Pregnant or lactating woman
* Minor
* Impossibility of signing consent
* No affiliation to a social security scheme (beneficiary or beneficiary)
* Person in emergency,
* Person of legal age subject to a legal protection measure (major under guardianship, guardianship or court order), or unable to express his or her consent
* Patient with at least 2 generalized tonic-clonic seizures per month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Numbers of crisis at baseline | 6 weeks
  The monthly frequency of crisis
Numbers of crisis under treatment | 5 weeks
  The monthly frequency of crisis during treatment period

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, Study Director — APHM
Locations (2):
- France (2):
  - Assistance Publique Des Hopitaux de Marseille, Marseille, PACA
  - Department of Epileptology and Cerebral Rhythmology, Hôpital La Timone, APHM, Marseille